CLINICAL TRIAL: NCT05874323
Title: The Relationship of RAGE Gene Polymorphism (rs1800625) With Type I Diabetes Mellitus Incidence, Severity, and Inflammatory Reactions in Egyptian Patients on MicroRNAs (MiRNA-34, MiRNA-146): A Case-control Study
Brief Title: The Relationship of RAGE Gene Polymorphism With Type I Diabetes in Egyptian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assistant professor, Future University in Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IDE00296
Record Dates: First submitted 2023-05-13; First posted 2023-05-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type I Diabetes Mellitus (Experimental): 177 patients with Type I Diabetes Mellitus
  Interventions: Genetic: Detection of RAGE gene polymorphism (rs1800625)
- Control (Other): include 177 Healthy Control Cases.
  Interventions: Genetic: Detection of RAGE gene polymorphism (rs1800625)

INTERVENTIONS:
Genetic: Detection of RAGE gene polymorphism (rs1800625) — Detection of RAGE gene polymorphism (rs1800625) By Molecular analysis (real time PCR)

SUMMARY:
Type I Diabetes Mellitus (TIDM) is a chronic metabolic disorder caused by the immune-mediated T-cell and macrophages that typically affects insulin-producing β-cells of Langerhans leading to cell destruction and absolute insulin deficiency. This study aimed to investigate the correlation of RAGE gene polymorphism rs1800625 with the incidence of type I diabetes mellitus in the Egyptian patients with the activity and the severity of the disease and to assess their association with inflammatory reactions in TIDM patients (IL-6, TNF-α). Also, this study investigated the relation between MiRNA-34, MiRNA-146, to TID severity and activity

DETAILED DESCRIPTION:
Type I diabetes mellitus (TIDM) is also called autoimmune diabetes, juvenile-onset or insulin-dependent diabetes mellitus . It is representing 10% of diabetes cases, estimated that most of these patients are less than 15 years old. The pathophysiology of TIDM is a complex and available data proposed the important cause for this disease such as autoimmune disease and some genetic factors TIDM is a chronic disease caused by the immune-mediated T-cell and macrophages attack on insulin-producing β-cells of Langerhans leading to cell destruction and absolute insulin deficiency. This will produce high blood sugar (hyperglycemia) and change in the proteins and lipids metabolism TIDM is usually characterized by the presence of anti-glutamic acid decarboxylase, islet of β-cell or insulin antibodies which identify the autoimmune processes, leads to β-cell destruction .

Type I diabetes mellitus is account for only a minority of the total burden of diabetes in a population, however it is considered the major type of diabetes in younger age .

Treatment of TIDM is more complex than other types of diabetes, as it cannot be regulated only by dietary interventions, as it is usually accompanied by severe complications, and has extreme variability due to the diverse ages of diagnosis. Primary treatment for TIDM include immune-suppressive drugs and continuous exogenous insulin that cover the primary pathophysiology of TIDM Currently, diabetes mellitus is diagnosed when hemoglobin A1C (HbA1c) is ≥6.5% or fasting plasma glucose (FPG) is ≥ 126 mg/dl or 2 hour postprandial plasma glucose is ≥ 200 mg/dl during an oral glucose tolerance test or a random plasma glucose is ≥ 200 mg/dl plus symptoms of diabetes .

Advanced glycation end products (AGEs) Advanced glycation end products (AGEs) are defined as a heterogeneous group of irreversibly reactive derivatives. They are formed by non-enzymatic glycation with tissue proteins, and shown to accumulate on long-lived proteins in diabetes mellitus . They generate oxidative stress and induce inflammation and they have been tied to be a factor in the development an unfavorable pro-inflammatory state implicated in many degenerative diseases, such as autoimmune diseases, diabetes, atherosclerosis, chronic renal failure, metabolic syndrome and its complications, and neurological diseases such as Alzheimer's disease, cardiovascular diseases (Kuzan and Aleksandra 2021). These harmful compounds can affect every type of cell in the body and are thought to be one factor in some age-related chronic diseases. Receptor for advanced glycation end products (RAGE) is a multi-ligand cell surface receptor that belongs to the immunoglobulin superfamily. RAGE activation by various ligands have been reported to induce LDL deposition, resulting in foam cell formation . Furthermore, it increase oxidative stress generation and subsequently increase inflammatory, proliferative, angiogenic, fibrotic, thrombogenic, and apoptotic reactions in numerous cell types via activation of many intracellular signaling pathways such as nuclear factor-κB (NF-κB) . RAGE expression is usually low in the majority of healthy adult tissues, but its levels are elevated under pathological conditions such as diabetes .

RAGE is a highly polymorphic gene, with around ten polymorphisms being predominantly studied. The genetic variations of RAGE should be considered as responsible for the development of many diseases (Serveaux et al., 2019). In addition, combining RAGE-circulating protein levels and RAGE polymorphisms may be used as a useful clinical tool to predict risk of vascular diseases. Indeed, sRAGE could be a valuable biomarker in many pathological states. It increases in patients with decreased renal function, and decreases in diabetic complications and coronary artery disease, but also elevated levels of sRAGE are often associated with end-stage disease . The genetic background of RAGE demonstrated that some gene polymorphisms are implicated in various pathological states, for example, diabetes complications, amplification of the inflammatory response, gastric cancer, and breast cancer . Recently, five main RAGE polymorphisms described (rs2070600, rs1800624, rs184003, and a 63 bp deletion) were not associated with either type 1 or type 2 diabetes . In this study, we focused on the principal RAGE polymorphism (rs1800625) and their potential pathological effect depending on the study of the Egyptian population with TIDM.

Rs1800625 Polymorphism The rs1800625 SNP (- 429 T > C) located in the upstream region and was found to increase the transcription of RAGE around twofold in vitro and so increase the RAGE expression, which might influence the pathogenesis of many diseases such as autoimmune and inflammatory diseases (Ahuja el al., 2022). In the presence of rs1800625 polymorphism, it is not only a higher expression of sRAGE but also, there is an increase of AGEs. Studies on different pathologies (inflammatory disease, cancer, coronary artery disease, lung disease, and myocardial infarction) focused on rs1800625, but with conflicting results. However the rs1800625 SNP was studied in different types of cancer but founded to be not involved in the pathogenesis of pancreatic cancer like RAGE is implicated There were numerous studies of SNP rs1800625 in diabetic patients, but with conflicting results. The rs1800625 SNP was significantly increased in type 2 diabetes subjects with retinopathy, compared to those without . Many studies demonstrated a correlation between rs1800625 polymorphism and diabetic complications. The rs1800625 and rs3134940 were founded to be increase (+65%) the risk of developing diabetic nephropathy and was associated with its early onset. The rs1800625 SNP was also associated with the development of insulin resistance, and in a Brazilian population there was a two-fold increase in the incidence of rs1800625 when subjects were diabetic. An analysis in infants with type I diabetes from the Finn Diane cohort reported that rs1800625 was more prevalent in type I diabetic patients than in controls . In diabetic subjects, rs1800625 was associated with higher HbA1c levels, with an increased incidence of type 1 diabetes.

The association of rs1800625 with cardiovascular risk has been evaluated, with again controversial results. The rs1800625 was associated with higher levels of circulating form of (RAGE) and an increased risk of developing coronary artery disease, especially in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* <18 Years

Exclusion Criteria:

* > 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
correlation of RAGE gene polymorphism rs1800625 with the incidence of type I diabetes | 4 months
  correlation of RAGE gene polymorphism rs1800625 with the incidence of type I diabetes using the TaqMan genotyping assay in the study population. Tumor necrosis factor-alpha (TNF-α), interleukin (IL-6) serum levels, and clinical parameters were measured using the enzyme-linked immunosorbent assay (ELISA) technique.

SECONDARY OUTCOMES:
the relation between MiRNA-34, MiRNA-146, to TID severity and activity. | 4 months
  the relation between MiRNA-34, MiRNA-146, to TID severity and activity. 146 were determined using quantitative real-time PCR (qPCR)

CONTACTS AND LOCATIONS:
Overall Officials: Amal mohamed, professor, Study Director — national hepatology and Tropical medicine institute
Locations (1):
- National Institute of Diabetes and Endocrinology's, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No